CLINICAL TRIAL: NCT01164332
Title: Investigation of the Sensitivity of Different Methods to Detect NRL972 in Healthy Volunteers During and After a 2-hour Intravenous Infusion of 10 and 30mg NRL972
Brief Title: Sensitivity of Alternative NRL972 Detection Methods in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Norgine (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: NRL972-01/2010 (AMET)
Record Dates: First submitted 2010-07-13; First posted 2010-07-16 (Estimated); Last update posted 2015-06-10 (Estimated); Status verified 2011-07

CONDITIONS: Cirrhosis
MeSH Terms: conditions — Fibrosis | interventions — NRL972

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Method A (Other): First experimental detection method
  Interventions: Other: NRL972
- Method B (Other): Second experimental detection method
  Interventions: Other: NRL972

INTERVENTIONS:
Other: NRL972 — Two-hour intravenous infusion of 5 and 15 mg per hour

SUMMARY:
The disposition of NRL972 after a 15-second intravenous injection of 2 mg NRL972 is distinctly slower in patients with hepatic cirrhosis and acute hepatitis than in healthy control subjects. NRL972 appears to be a suitable investigational marker of hepatic transporter clearance dysfunction.

Although the pharmacokinetics of NRL972 provide a reliable differentiation between subject groups, this approach relies on precisely timed sampling of venous blood, cautious preparation, handling and on-site storage of plasma samples, the transfer of samples to a central laboratory for analysis, and the availability of a validated assay procedure.

For these reasons, there is interest in developing and validating alternative methods for determining the concentration of NRL972 in venous blood. Two such methods have been developed to date, but their utility in determining NRL972 pharmacokinetics has yet to be established.

ELIGIBILITY:
Inclusion Criteria:

Subjects meeting the following conditions will be eligible for enrolment:

* Males or females (females of non-childbearing potential or of childbearing potential while taking medically appropriate contraception)
* Caucasian
* Age: 20 to 45 years
* BMI 20 - 26 kg.m-2
* Healthy based on the pre-study examination
* Suitable veins for easy cannulation
* Willing and able to provide informed consent

Exclusion Criteria:

Subjects of any of the following categories will be excluded from enrolment:

General - all subjects

* Previous participation in the trial
* Participant in any other trial during the last 90 days
* Donation of blood during the last 60 days or a history of blood loss exceeding 300 mL within the last 3 months
* History of any clinically relevant allergy
* Presence of any acute or chronic infection
* Presence or history of any relevant co-morbidity
* Resting systolic blood pressure > 160 or < 90 mmHg, diastolic blood pressure > 95 or < 50 mmHg
* Clinically relevant ECG-abnormalities, prolonged QTc with > 450 msec in males and > 460 msec in females in particular
* Presence of any relevant abnormality in the laboratory safety tests, especially low haemoglobin, increased liver enzymes
* Positive serology for HBsAg, anti HBc and anti HCV
* Positive HIV test
* Positive alcohol or urine drug test on recruitment
* History of alcohol and/or drug abuse and/or daily use of > 30 g alcohol
* Smoking more than 10 cigarettes/day or equivalent of other tobacco products
* Use of prohibited medication
* Suspicion or evidence that the subject is not trustworthy and reliable
* Suspicion or evidence that the subject is not able to make a free consent or to understand the information in this regard

General - all females

* Positive pregnancy test
* Lactating
* Not using appropriate contraception in premenopausal women

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2010-07; Primary Completion 2010-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Ratios of the plasma concentration at 30 minutes post-infusion to the concentrations at 10 and 15 minutes post-infusion | Up to 4 hours post-dose

SECONDARY OUTCOMES:
Adverse events | Up to 4 hours post-dose
Vital signs | Up to 4 hours post-dose
ECG | Up to 4 hours post-dose
Clinical laboratory blood tests | Up to 4 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Eva Peterfai, MD, Principal Investigator — Drug Research Center Ltd.
Locations (1):
- Phase I-II study clinical of the Drug Research Center Ltd., Balatonfüred, Hungary